CLINICAL TRIAL: NCT04389944
Title: Amotosalen-Ultraviolet A Pathogen-Inactivated Convalescent Plasma in Addition to Best Supportive Care and Antiviral Therapy on Clinical Deterioration in Adults Presenting With Moderate to Severe Coronavirus Disease 2019 Infectious Disease (COVID-19)
Brief Title: Amotosalen-Ultraviolet A Pathogen-Inactivated Convalescent Plasma in Addition to Best Supportive Care and Antiviral Therapy on Clinical Deterioration in Adults Presenting With Moderate to Severe COVID-19
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Basel, Switzerland (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Req-2020-00508; me20khanna2
Record Dates: First submitted 2020-05-12; First posted 2020-05-15 (Actual); Last update posted 2020-08-04 (Actual); Status verified 2020-08

CONDITIONS: Coronavirus Disease 2019 Infectious Disease (COVID-19 Infection)
Keywords: convalescent plasma; Severe Acute Respiratory Syndrome Coronavirus 2 (SARS-CoV-2)
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- convalescent plasma treatment (Experimental): After confirmation of negative SARS-CoV-2 polymerase chain reaction (PCR) in two consecutive nasal swabs or 28 days after resolution of symptoms, donor check is performed and plasma donation occurs by apheresis. The plasma is photochemically pathogen reduced using the INTERCEPT Blood System.
  In addition to standard of care, SARS-CoV-2 infected patients for whom blood group compatible convalescent plasma is available and who are willing to sign the informed consent receive convalescent plasma as follows: 200ml at enrolment and 200ml at 12-24 hours follow-up.
  Interventions: Other: convalescent plasma application to SARS-CoV-2 infected patients

INTERVENTIONS:
Other: convalescent plasma application to SARS-CoV-2 infected patients — In addition to standard of care, SARS-CoV-2 infected patients for whom blood group compatible convalescent plasma is available and who are willing to sign the informed consent receive convalescent plasma as follows: 200ml at enrolment and 200ml at 12-24 hours follow-up.

SUMMARY:
This project investigates individual treatments using convalescent severe acute respiratory Syndrome Coronavirus 2 (SARS-CoV-2) plasma in SARS-CoV-2 infected patients at risk for disease progression. In addition to standard of care, SARS-CoV-2 infected patients for whom blood group compatible convalescent plasma is available and who are willing to sign the informed consent receive convalescent plasma. Only patients with moderate to severe disease at risk for transfer to intensive care unit or patients at the intensive care unit with limited treatment options will be treated.

ELIGIBILITY:
Inclusion Criteria for donors:

* male patients who have been tested positive for SARS-CoV2 at University Hospital Basel, Switzerland or in the near surroundings more than 10 days before enrolment
* 18-60 years of age
* asymptomatic (thus successfully overcome COVID-19) >14 days back
* two consecutive naso-pharyngeal swabs tested negative for quantitative PCR-test for SARS-CoV-2 prior to plasma donation to demonstrate infection Resolution, or more than 28 days asymptomatic after SARS-CoV2 infection
* Body weight of at least 50 kg
* donor eligibility criteria according to the Swiss Red Cross Blood Transfusion Service as for regular blood donation

Exclusion Criteria for donors:

* Female donors are excluded from plasma donation
* Treatment with Actemra® (Tocilizumab) in the course of COVID-19
* Current hospitalization
* Current or previous relevant medical conditions that pose a risk for the donor

Inclusion Criteria for COVID-19 infected patients:

* SARS-CoV-2 infection confirmed by PCR in respiratory secretions (naso- pharyngeal swab, broncho-alveolar lavage, sputum)
* hospitalized
* pulmonary infiltrates compatible with COVID-19 on CT-scan
* availability of blood group compatible convalescent plasma
* signed informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2020-03-31 (Actual); Primary Completion 2020-06-30 (Actual); Study Completion 2020-06-30 (Actual)

PRIMARY OUTCOMES:
Serious adverse events in convalescent plasma treated patients | From baseline (enrolment) to 24 hours follow-up
  Serious adverse events during the study period include transfusion reaction (fever, rash), transfusion related acute lung injury (TRAU) , transfusion associated circulatory overload (TACO) , transfusion related infection
Virologic clearance in nasopharyngeal swab of convalescent plasma treated patients | at Baseline (admission to Covid-ward), day -1 (before plasma), day 1 (after plasma), day7, day 14, day 28
  Change in SARS-CoV2 quantitative in nasopharyngeal swab
Transfer to ICU | at Baseline (admission to Covid-ward) until day 28
  Transfer to ICU
in-hospital death | at Baseline (admission to Covid-ward) until day 28
  in-hospital death
Virologic clearance in plasma of convalescent plasma treated patients | at Baseline (admission to Covid-ward), day -1 (before plasma), day 1 (after plasma), day7, day 14, day 28
  Change in SARS-CoV2 quantitative in plasma

SECONDARY OUTCOMES:
Time to discharge from hospital after enrolment | at Baseline (admission to Covid-ward) until discharge (approx. 28 days)
  Duration of hospitalisation
Humoral immune response | at Baseline (admission to Covid-ward), day -1 (before plasma), day 1 (after plasma), day7, day 14, day 28
  Rise of SARS-CoV-2 antibody titers (on day 1, 7, 14 and 28)

CONTACTS AND LOCATIONS:
Overall Officials: Andreas Buser, Prof. Dr. med., Principal Investigator — Blutspendezentrum SRK beider Basel, Universitätsspital Basel
Locations (1):
- Blutspendezentrum SRK beider Basel, University Hospital Basel, Basel, Switzerland